CLINICAL TRIAL: NCT05857475
Title: Efficacy of CPAP Therapy on Pulmonary Function Test in Patients With COPD-OSA Overlap Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MahidolU 4564
Record Dates: First submitted 2023-03-03; First posted 2023-05-12 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: COPD; OSA; Lung Function Decreased
Keywords: COPD-OSA overlap syndrome; Pulmonary function test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: To compare pulmonary function of COPD-OSA overlap subjects who using and not using (waiting list for PAP therapy) in the period of 2 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP therapy (Experimental): CPAP therapy will be used in this arm for 2 month.
  Interventions: Device: CPAP therapy
- Control (Other): CPAP therapy will not be used in this arm for 2 month. (subject were assign to normal waiting list in order to borrowing hospital PAP machine.)
  Interventions: Other: Control

INTERVENTIONS:
Device: CPAP therapy — Continous positive airway pressure therapy
  Arms: CPAP therapy
Other: Control — No CPAP
  Arms: Control

SUMMARY:
To evaluate efficacy of CPAP Therapy on Pulmonary Function Test in Patients With COPD-OSA Overlap Syndrome

DETAILED DESCRIPTION:
To evaluate efficacy of CPAP Therapy on Pulmonary Function Test in Patients With COPD-OSA Overlap Syndrome by 6 minute walking distance and oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with COPD by GOLD guideline criteria (Post bronchodilator FEV1/FVC < 0.7 or < LLN) with post bronchodilator FEV1 = 30-80%
* Diagnosis with obstructive sleep apnea with AHI > 15 event/hr. (Moderate OSA or more)
* Age between 40-80 years
* Stable disease prior to inclusion.

Exclusion Criteria:

* Diagnosis with > 50% of central sleep apnea event
* History of COPD exacerbation during the past 8 week prior to inclusion.
* Subjects who cannot perform spirometry test or walking test
* Subjects with recording history of chronic heart failure, significant arrhythmias, acute myocardial infarction, moderate to severe mitral or aortic valve disease and pulmonary hypertension.
* Subjects with interstitial lung disease.
* Subjects with neuromuscular disease.
* Subjects with morbid obesity (BMI >/=35)
* Subjects with chronic respiratory infection.
* Subjects with chronic CO2 retension (PaCO2 >/= 45 from arterial blood gas analysis) or Transcutaneous CO2 during sleep test >/= 45 or Serum bicarbonate level > 27
* Subjects with acute or active respiratory infecton during 2 week prior to inclusion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
6 minute walking test distance | 2 months
  To measure distance subject could walk during the period of 6 minute

SECONDARY OUTCOMES:
Quality of life by questionaires: COPD Assessment Test (CAT) | 2 months
  Using COPD Assessment Test (CAT) questionaires to assessing globally the impact of COPD (cough, sputum, dyspnea, chest tightness, activities, confident, sleep and sleep) on health status
  - Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life
Quality of life by questionaires: modified British Medical Research Council Dyspnea Scale (mMRC) | 2 months
  Using COPD modified British Medical Research Council Dyspnea Scale (mMRC) to assess the degree of functional disability due to dyspnea.
Quality of life by questionaires: St. George's Respiratory Questionnaire (SGRQ) | 2 months
  Using St. George's Respiratory Questionnaire (SGRQ) to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.
  SGRQ is divided into 2 part
  * Part I (Symptoms): several scales.
  * Part II (Activity and Impacts): dichotomous (true/false). Scores range from 0 to 100, with higher scores indicating more limitations.
Quality of life by Sleep quality questionaires: Pittsburgh Sleep Quality Index (PSQI) | 2 months
  Using Pittsburgh Sleep Quality Index (PSQI) to assesses adult patients' sleep quality and disturbances over one month with question about Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Quality of life by Sleep quality questionaires: Functional Outcomes of Sleep Questionnaire (FOSQ) | 2 months
  Using Functional Outcomes of Sleep Questionnaire (FOSQ) to to determine functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment.
  The questionaire ask about activity level, vigilance, intimacy and sexual relationships, general productivity, social outcome, rate the difficulty of performing a given activity on a 4-point scale (no difficulty to extreme difficulty)
Quality of life by Sleep quality questionaires: Epworth Sleepiness Scale (ESS) | 2 months
  Using Epworth Sleepiness Scale (ESS) to measure sleepiness in daily life. The ESS asks the patient to rate their likelihood of falling asleep under 8 different circumstances.
Quality of life by Sleep quality questionaires: Lausanne NoSAS (Neck circumference, Obesity, Snoring, Age, Sex) score | 2 months
  Using Lausanne NoSAS (Neck circumference, Obesity, Snoring, Age, Sex) score to guide identification of individuals at risk of sleep-disordered breathing
Aerobic capacity | 2 months
  Measure oxygen consumption during performing 6 minute walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided